CLINICAL TRIAL: NCT02795520
Title: Phase I/II and Pharmacological Study of Intravenous OTS167 in Patients With Refractory or Relapsed Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, Advanced Myelodysplastic Syndromes, Advanced Myeloproliferative Neoplastic Disorders, or Advanced Chronic Myelogenous Leukemia
Brief Title: Pharmacological Study of Intravenous OTS167 in Patients With Refractory or Relapsed Acute Myeloid Leukemia, Acute Lymphoblastic Leukemia, Advanced Myelodysplastic Syndromes, Advanced Myeloproliferative Neoplastic Disorders, or Advanced Chronic Myelogenous Leukemia
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: slow patient accrual
Sponsor: OncoTherapy Science, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: OTS167-SE02
Record Dates: First submitted 2016-05-06; First posted 2016-06-10 (Estimated); Last update posted 2021-11-24 (Actual); Status verified 2021-11

CONDITIONS: AML; Advanced MDS; ALL; Advanced CML; Advanced MPNs

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- OTS167IV (Experimental)
  Interventions: Drug: OTS167IV

INTERVENTIONS:
Drug: OTS167IV

SUMMARY:
The purpose of Phase I of this study is to test the safety and tolerability of the investigational drug, OTS167, and that of Phase II of this study is to confirm the potential response benefit of OTS167.

OTS167 is a maternal embryonic leucine zipper kinase (MELK) inhibitor which demonstrated antitumor properties in laboratory tests. It is being developed as an anti-cancer drug. In this study OTS167 will be administrated to patients with AML, ALL, advanced MDSs, advanced MPNs, or advanced CML.

ELIGIBILITY:
Inclusion Criteria:

1. Diagnosis of:

   * Relapsed or refractory AML (refractory to a standard anthracycline-based induction regimen or a hypomethylating agent for patients unfit for intensive chemotherapy or for whom no standard or curative therapy exists),
   * ALL,
   * Acute biphenotypic leukemia (assigned to the appropriate group by the treating physician by documented analysis of relevant laboratory values and pathology/cytogenetics),
   * Advanced MDS defined as ≥5% bone marrow blasts or ≥2% blasts in the peripheral blood (including patients who have progressed following treatment with hypomethylating agents),
   * Advanced MPN (excluding patients with ET, PV, or low risk MF), and MDS/MPN overlap syndrome with ≥5% bone marrow blasts or ≥2% blasts in the peripheral blood, or
   * Advanced CML after failure/progression of at least 3 prior TKIs
2. Age ≥18 years
3. No prior antineoplastic drug therapy for at least 14 days, with the exception of hydroxyurea, prior to starting OTS167. Patients with rapidly proliferative disease may continue to receive hydroxyurea
4. Patients refractory to all approved therapies or for which no approved or conventional therapies are available
5. Patients with a diagnosis of advanced CML must have been treated with 3 prior TKIs, and the last therapy must have been discontinued at least 14 days prior to starting OTS167
6. Adequate organ function as defined below:

   * Liver function (total bilirubin <2 mg/dL and aspartate aminotransferase and/or alanine aminotransferase <3 × upper limit of normal (ULN) or <5 × ULN if related to leukemic involvement)
   * Renal function (creatinine <1.5 × ULN)
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 2
8. Negative urine pregnancy test within 1 week prior to Cycle 1 Day 1 for each woman of childbearing potential
9. Able to understand the potential risks, benefits, and requirements of the study and are willing to provide informed consent; an informed consent form (ICF) for this study that is signed by the patient or his/her legally authorized representative is required prior to enrollment

Exclusion Criteria:

1. Pregnant or breastfeeding patients (pregnant and breastfeeding women are excluded from this study because the agents used in this study may have unknown or unrecognized potential for teratogenic or abortifacient effects). Patients of childbearing potential must consent and agree to practice documented (type) adequate contraception during the course of on study treatment.
2. Evidence of any form of active, uncontrolled, bacterial, viral (including hepatitis A, B, or C or known human immunodeficiency virus [HIV] seropositivity), or fungal infection. Patients who are positive for hepatitis B core antibody, hepatitis B surface antigen, or hepatitis C antibody must have a negative polymerase chain reaction (PCR) result before enrollment; those who are PCR-positive will be excluded. Evidence of congestive heart failure (New York Heart Association Class III or IV); myocardial infarction or stroke within 6 months; unstable angina; uncontrolled or unstable/medically important cardiac arrhythmia; prolonged QT interval corrected for heart rate (QTc) >450 msec (males) or >470 msec (females); uncontrolled epilepsy; uncontrolled bleeding; recent major surgical procedures within 30 days before Cycle 1 Day 1 without full recovery from the same; or any other serious comorbid medical condition that would preclude investigational study treatment
3. Any psychiatric illness/social situations that would limit compliance with study requirements
4. Documented hypersensitivity to any of the components of OTS167 or supportive care medicaments
5. Central nervous system (CNS) leukemia
6. MPN patients with ET, PV, or low risk MF
7. Women of childbearing potential and men must agree prior to study entry to use appropriate contraception for the duration of study participation and until 30 days after receipt of the last dose of study drug
8. Documented concurrent malignancy. Exceptions include cervical carcinoma in-situ, non-melanoma skin cancer (basal and squamous cell carcinoma), localized prostate cancer (Gleason score <6), and resected melanoma-in-situ. Other localized solid tumors in situ and other low risk cancers may also be exempt after discussion with the Sponsor Medical Monitor.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2021-05 (Actual); Study Completion 2021-09 (Actual)

PRIMARY OUTCOMES:
Adverse events assessed by CTCAE v4.03 | Up to 30 days after last dose of study drug

CONTACTS AND LOCATIONS:
Overall Officials: Olatoyosi Odenike, MBBS, Principal Investigator — University of Chicago, Ilinois
Locations (2):
- United States (2):
  - University of Chicago, Chicago, Illinois
  - Weill Cornell Medicine, New York, New York